CLINICAL TRIAL: NCT05051644
Title: An Adaptive Walking Intervention to Manage Chronic Pain in Veterans With Opioid Use Disorder Engaged in Opioid Agonist Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NURP-001-21S; IK2CX002286 (NIH)
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder; Chronic Pain
Keywords: Chronic Pain; Opioid Use Disorder; opioid agonist treatment; medications for opioid use disorder; methadone; buprenorphine; walking; exercise
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Recruitment strategies will week to minimize the amount of time between screening visit and treatment start date. After completing screening visit, Veterans will begin a 7 day baseline EMA run-in period leading up to the start of the treatment week. First treatment session will be scheduled 7 days after screening visit. The feasibility of these procedures will be evaluated in Aim 1. Veterans who provide pedometer and EMA survey data on at least 3 days during baseline EMA will be randomized. Veterans will be randomized to either S2C or control in a 1:1 ratio using permuted block randomization stratified by OAT type (1=buprenorphine, 2=methadone) and sex (1=male, 2=female). A variable block size of 2 and 4 will be used to maintain balanced assignment to condition.
Who Masked: Participant, Outcomes Assessor
Masking Description: General terms will be used when recruiting potential participants and in the informed consent. Study title on informed consent and recruitment materials will be "Enhancing self-management skills for individuals with opioid use disorder." Study measures (both in clinic and EMA) will be described as collecting data on problems that Veterans with OUD commonly report (e.g., negative mood, pain, quality of life, stress, etc.) and may improve with increased engagement in treatment. All in person assessment for post-treatment, 3 month follow up, and 6 month follow up will be collected by a research staff member who is blind to study condition. Data from EMA surveys at each time point will be provided by study participant whom is already blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steps 2 Change (S2C) (Experimental): Participants randomized to S2C will be scheduled for 30-45 minute weekly treatment sessions held over four consecutive weeks in the outpatient OAT clinic. Veterans will be expected to increase their average step counts by 10% over their prior week's average. Session 1 will provide pain education including a discussion the biopsychosocial treatment model for chronic pain and benefits of activity. Session 2 and 3 will emphasize benefits of low impact physical activity and introduce activity pacing to address pain related to cycles of over activity and subsequent sedentary behavior. Session 4 will help develop a treatment plan to continue walking and identify possible barriers to meeting goals.
  Interventions: Behavioral: Steps 2 Change (S2C)
- Control (Active Comparator): Participants randomized to control will be scheduled for 30-45 minute weekly treatment sessions held over four consecutive weeks focused on problems associated with MOUD, substance use, and general self-management strategies. Importantly, group will explicitly avoid talking about pain coping skills and setting goals for daily step targets.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Steps 2 Change (S2C) — Session 1 will provide pain education including a discussion the biopsychosocial treatment model for chronic pain. Session 2 and 3 will introduce a progressive walking program with individual goals and weekly step count benchmarks and introduce activity pacing to address pain flare ups caused by cycles of over activity and subsequent sedentary behavior. Veterans will be expected to increase their average step counts by 10% over their prior week's average starting in Session 2. Session 4 will help develop a treatment plan to continue walking and identify possible barriers to meeting goals.
  Arms: Steps 2 Change (S2C)
Behavioral: Control — The control will be matched for treatment exposure and individual attention. Treatment discussion will explicitly avoid problems associated with MOUD, substance use, and general self-management strategies. Importantly, group will explicitly avoid talking about pain coping skills and setting goals for daily step targets.
  Arms: Control

SUMMARY:
Severe chronic pain and opioid use disorder (OUD) occur at significantly higher rates in Veterans compared to the general population. Chronic pain often persists despite engagement in opioid agonist treatment (OAT), the first line treatment for OUD. Recent VA guidelines strongly recommend non-pharmacologic treatment for chronic pain, but individuals with OUD are frequently excluded from pain treatment studies. There is a need for evidence-based pain treatments that compliment OAT for Veterans with chronic pain and OUD. In this study, the investigators will determine feasibility and acceptability for a behaviorally focused pain treatment that includes pain education and a pedometer assisted adaptive walking program for Veterans receiving OAT for OUD. Potential treatment outcomes will be repeatedly assessed using a mobile device, and study-provided pedometers. By offering pain treatment within OAT clinical care, the investigators hope to decrease stigma and increase access for Veterans with chronic pain and OUD.

DETAILED DESCRIPTION:
The proposed study will address the pain treatment knowledge gap in Veterans with opioid use disorder (OUD) by piloting a behaviorally-based walking pain treatment for Veterans with chronic pain and OUD. Steps to Change (S2C) is a pain-focused treatment comprised of brief weekly 30-45-minute treatment sessions held over four consecutive weeks within the a Veterans Health Administration opioid agonist treatment (OAT) clinic. To date, no study has evaluated a pedometer-assisted walking program in individuals with chronic pain and OUD engaged in OAT. Topics for S2C include biopsychosocial pain education, pacing activities, benefits of physical activity, and an adaptive walking program derived from Cognitive Behavioral Therapy for chronic pain (CBT-CP) modules. The control will be matched for treatment exposure and attention. Veterans in both conditions will be provided a pedometer to record daily step counts as an objective measure of physical activity. Importantly, pain is a dynamic process that is known to vary over time and context. Veterans in both conditions will complete ecological momentary assessment (EMA) surveys, where behavior is repeatedly sampled using a mobile device.

The study objectives align closely with the description of a Stage IB pilot trial. Stage IB research determines feasibility and pilot testing of an adaptation or refinement of an existing intervention. Walking is a core component of CBT-CP and physical activity has a strong evidence base as a pain treatment for individuals with chronic pain; however, a walking program for chronic pain has not been evaluated in Veterans with chronic pain and OUD receiving OAT. Aim 1 will determine feasibility of study procedures including randomization, retention, fidelity, and proposed study outcomes of S2C and control conditions. Evaluating the feasibility of treatment and best practices for how quickly Veterans can be screened, consented, and randomized to start treatment is a critical step to inform a larger Stage II efficacy trial. In addition, the investigators will evaluate treatment attendance and retention in both S2C and control conditions to determine feasibility as well as discrimination of conditions for fidelity. The investigators will also collect data on mobile phone ownership and compare EMA survey response rates between conditions to inform future efficacy studies. The investigators expect that treatment attendance, retention, and survey responses for S2C will be equal to or superior then control. Aim 2 will establish acceptability of S2C and health education control by assessing intervention credibility and satisfaction at post-treatment. The investigators expect that Veterans in both conditions will report treatment as credible and satisfying. Finally, Aim 3 will evaluate preliminary evidence for whether S2C, compared to control, reduces pain interference assessed via interference items on the PEG. Primary endpoint will be at post-treatment, but the investigators will also evaluate durability or sleeper effects on pain interference at 3- and 6-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM5 criteria for OUD and receiving stable (i.e., unchanged in 2 weeks) dose of OAT (i.e., buprenorphine or methadone) in VACHS outpatient addiction clinic
* Report high impact or bothersome chronic pain defined by experiencing pain on most days or every day in the past 3 months that limits general activity or enjoyment
* Self-reported ability to walk 1 block
* Access to a mobile phone with active data plan

Exclusion Criteria:

* Untreated major psychiatric disorders (e.g., bipolar disorder, psychotic disorder)
* Current (i.e., past month) active suicidal ideation
* Substance use disorder requiring inpatient detoxification
* Currently engaged in CBT for chronic pain treatment
* Planned surgical intervention for pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Ross MacLean, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that underlies published reported results after deidentification (text, tables, figures, appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 months to 36 months after publication of primary findings.
Access Criteria: Up to 36 months after publication of primary findings, de-identified data can only be used for research purposes with a priori hypotheses including secondary analyses and/or meta-analysis combined with other datasets. Proposals should be directed to robert.maclean@va.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veteran participants were recruited to the study in several ways, including: (1) hanging study flyers in outpatient clinics, (2) study staff attending clinic team meetings to provide information about the study and invite Veteran referrals to the study coordinator; (3) mailing opt-out letters allowing Veterans engaged in outpatient OAT to be contacted via phone call or state they do not wish to participate.
Pre-assignment Details: After consent and screening visit, participants began 7-days of baseline mobile surveys including three random and one end of day survey per day (4 total). To be randomized, Veterans will need to complete at least 3 end of day surveys with complete step and pain interference data. If a Veteran fails to complete surveys in first 2 days of baseline EMA week, research staff will contact Veteran to assess for technical difficulties and encourage survey completion.
Groups:
- Steps 2 Change (S2C): Participants randomized to S2C will be scheduled for 30-45 minute weekly treatment sessions held over four consecutive weeks in the outpatient OAT clinic. Veterans will be expected to increase their average step counts by 10% over their prior week's average starting after Session 1. Session 1 will provide pain education including a discussion the biopsychosocial treatment model for chronic pain and benefits of activity. Session 2 and 3 will emphasize benefits of low impact physical activity and introduce activity pacing to address pain flare ups caused by cycles of over activity and subsequent sedentary behavior. Session 4 will help develop a treatment plan to continue walking and identify possible barriers to meeting goals.
- Control: Participants randomized to control will be scheduled for 30-45 minute weekly treatment sessions held over four consecutive weeks focused on problems associated with MOUD, substance use, and general self-management strategies. Importantly, group will explicitly avoid talking about pain coping skills and setting goals for daily step targets. The control will be matched for treatment exposure and individual attention.
Period: Overall Study
Arm/Group | Steps 2 Change (S2C) | Control
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steps 2 Change (S2C) | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.7) | 54.4 (11.4) | 53.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 28 | 27 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 19 | 24 | 43
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
OAT type [Count of Participants; unit: Participants]
  Buprenorphine | 19 | 19 | 38
  Methadone | 11 | 11 | 22
Length of time on current OAT [Mean (Standard Deviation); unit: years] | 6.0 (4.8) | 5.2 (4.1) | 5.5 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Treatment retention measured as the number of attended sessions (0-4; higher number is better)
Time Frame: Up to 5 weeks
Measure: Mean (Standard Deviation); unit: number of sessions attended
Arm/Group | Steps 2 Change (S2C) | Control
Number analyzed (Participants) | 30 | 30
number of sessions attended | 3.7 (0.5) | 3.6 (0.9)

2. Primary Outcome: Acceptability
Description: Credibility measured using the Credibility/Expectancy Questionnaire with separate scores for credibility and expectancy (3-27; higher number is better).
Time Frame: After the first session, on the same calendar day
Population: Credibility survey was not completed by 6 participants (3 in each group).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Steps 2 Change (S2C) | Control
Number analyzed (Participants) | 27 | 27
Score on a scale
  Credibility | 18.7 (4.4) | 20.2 (4.6)
  Expectancy | 15.7 (4.8) | 15.9 (5.8)

3. Primary Outcome: Fidelity
Description: Fidelity measured as clinician adherence and competence in delivering study interventions using the Yale Adherence and Competence System (1-5; higher number is better).
Time Frame: Up to 5 weeks
Population: We randomly selected 24 participants (12 in each arm) to evaluate fidelity using one of their session recordings.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Steps 2 Change (S2C) | Control
Number analyzed (Participants) | 12 | 12
Score on a scale | 3.1 (0.2) | 3.2 (0.2)

4. Secondary Outcome: Pain Interference
Description: Pain interference measured using the average difference from baseline to post-treatment of two interference items on the PEG3: "What number best describes how pain is interfering with your life?" and "What number best describes how pain is interfering with your general activity?" (0-10; lower number is better)
Time Frame: 0-5 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Steps 2 Change (S2C) | Control
Number analyzed (Participants) | 30 | 29
Units on a scale | 0.8 (2.1) | 0.9 (2.8)
Statistical Analysis 1: Comparison: Steps 2 Change (S2C) vs Control; Test type: Other — The estimated mean changes from baseline to post-treatment, mean differences and 95% CI between groups at post-treatment; Mean change = 0.34, 95% CI 2-sided [-0.94 to 1.63]

5. Other Pre Specified Outcome: Pain Interference
Description: Pain interference measured using the average difference from baseline to follow-up of two interference items on the PEG3: "What number best describes how pain is interfering with your life?" and "What number best describes how pain is interfering with your general activity?" (0-10; lower number is better)
Time Frame: 3-month and 6-month follow up
Population: Missing data from participants who did not complete follow up visits.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Steps 2 Change (S2C) | Control
Number analyzed (Participants) | 30 | 29
Score on a scale
  3-month: number analyzed (Participants) | 27 | 24
  3-month | 1.0 (2.2) | 0.9 (3.0)
  6-month: number analyzed (Participants) | 23 | 24
  6-month | 1.2 (2.4) | 0.9 (2.8)
Statistical Analysis 1: Comparison: Steps 2 Change (S2C) vs Control; Test type: Other — The estimated mean changes from baseline to 3-months, mean differences and 95% CI between groups at 3-months; mean change = 0.03, 95% CI 2-sided [-1.05 to 1.5]
Statistical Analysis 2: Comparison: Steps 2 Change (S2C) vs Control; Test type: Other — The estimated mean changes from baseline to 6-months, mean differences and 95% CI between groups at 6-months; mean change = -0.11, 95% CI 2-sided [-1.6 to 1.4]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from screening through final follow up (i.e., 9-months).
Description: The investigators used definitions consistent with clinicaltrials.gov. Possible adverse events were collected by study clinicians inquiring
Groups:
- Steps 2 Change (S2C): Participants randomized to S2C will be scheduled for 60-minute weekly treatment sessions held over four consecutive weeks in the outpatient OAT clinic. Veterans will be expected to increase their average step counts by 10% over their prior week's average. Session 1 will provide pain education including a discussion the biopsychosocial treatment model for chronic pain and benefits of activity. Session 2 and 3 will emphasize benefits of low impact physical activity and introduce activity pacing to address pain related to cycles of over activity and subsequent sedentary behavior. Session 4 will help develop a treatment plan to continue walking and identify possible barriers to meeting goals.
  Steps 2 Change (S2C): Session 1 will provide pain education including a discussion the biopsychosocial treatment model for chronic pain. Session 2 and 3 will introduce a progressive walking program with individual goals and weekly step count benchmarks and introduce activity pacing to address pain flare ups caused by cycles of over activity and subsequent sedentary behavior. Veterans will be expected to increase their average step counts by 10% over their prior week's average starting in Session 2. Session 4 will help develop a treatment plan to continue walking and identify possible barriers to meeting goals.
- Control: Participants randomized to control will be scheduled for 60-minute weekly treatment sessions held over four consecutive weeks focused on problems associated with MOUD, substance use, and general self-management strategies. Importantly, group will explicitly avoid talking about pain coping skills and setting goals for daily step targets.
  Control: The control will be matched for treatment exposure and individual attention. Treatment discussion will explicitly avoid problems associated with MOUD, substance use, and general self-management strategies. Importantly, group will explicitly avoid talking about pain coping skills and setting goals for daily step targets.
Arm/Group | Steps 2 Change (S2C) | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 4/30
Other Adverse Events (participants affected / at risk) | 14/30 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steps 2 Change (S2C) (N=30) | Control (N=30)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Three day inpatient for psychological observation, participant self presented to PER for depression with +SI and plan to OD.
Drug Overdose (Psychiatric disorders) | 1 (1) | 2 (2) — Overdose of non-prescription opioids.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Admitted to MICU after presenting to ER with shortness of breath.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steps 2 Change (S2C) (N=30) | Control (N=30)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (11) | 6 (6) — Report of increased pain
Detox (Psychiatric disorders) | 2 (3) | 1 (1) — Presented to PER for drug or alcohol detox
Physical accident (Investigations) | 1 (1) | 1 (1) — Presented to medical ER for evaluation
Illness (Infections and infestations) | 5 (8) | 5 (5) — Presented to ER with symptoms of illness
Vision problems (Eye disorders) | 1 (1) | 1 (1) — Presented to clinic with blurred vision
Medication (Psychiatric disorders) | 1 (1) | 1 (1) — Presented to ER for medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT05051644/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05051644/ICF_000.pdf